CLINICAL TRIAL: NCT00271427
Title: Selenium Treatment in Autoimmune Thyroiditis: Long Term Follow-Up With Variable Doses
Brief Title: Selenium Treatment in Autoimmune Thyroiditis (AIT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STAIT
Record Dates: First submitted 2005-12-30; First posted 2006-01-02 (Estimated); Last update posted 2006-08-23 (Estimated); Status verified 2004-12

CONDITIONS: Autoimmune Thyroiditis; Hashimotos Thyroiditis
Keywords: Thyroiditis; Autoimmune; Hashimoto's; TPOAb; Selenium
MeSH Terms: conditions — Thyroiditis, Autoimmune; Thyroiditis | interventions — Selenium

INTERVENTIONS:
Drug: L-Selenomethionine

SUMMARY:
Selenium suppresses autoimmune destruction of thyrocytes and decreases titers of serum TPOAb in AIT patients. Older 4 clinical trials approved the efficacy of the daily dose of 200micg. It's believed that Se saturates the deficient stores of GPX so GPX saves the thyrocytes against to oxidative stresses. Although less than 70 micg/d is sufficient to maximize GPX activity, none of the authors tested the doses less than 200 micg/d. Our hypothesis was that If 100 micg/d can not suppress the TPOAb titers,it means autoimmune destruction can not be blocked by saturation of deficient stores of GPX solely and the mechanism of action requires more than repletion of deficient stores. It's important not only to estimate the optimal dose but to understand the mechanism of action. High dose therapy may also suppress TPOAb levels in Se-non-deficient AIT patients, if it is so, Se therapy may becomes the solely treatment modality which can suppress the autoimmunity in more than 400 million AIT patients. Because there've been no way to suppress autoimmune war and replacement of LT4 had been the only treatment modality for palliation. An other independent part of the study is to test the effect of Se in adolescent AIT patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically approved AIT patients who do not use any medication other than LT4 to keep TSH in the lower half of normal range.

Exclusion Criteria:

* Any kind of drug use other than LT4 or any kind of known pathology which may effect GIS absorption.

Ages: 15 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2004-12; Study Completion 2005-08

PRIMARY OUTCOMES:
statistically important change in serum TPOAb titers.

SECONDARY OUTCOMES:
Observe the long term effects to 9th mo.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Turker, Specialist, Principal Investigator — Dep. of Nuc. Med., Gulhane Military Academy of Medicine; Kamil Kumanlioglu, Prof., Study Director — Dep. of Nuc. Med., Ege University Faculty of Medicine.
Locations (1):
- Dep. of Nuc. Med., Ege University Faculty of Medicine., Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Turker O, Kumanlioglu K, Karapolat I, Dogan I. Selenium treatment in autoimmune thyroiditis: 9-month follow-up with variable doses. J Endocrinol. 2006 Jul;190(1):151-6. doi: 10.1677/joe.1.06661. PMID 16837619